CLINICAL TRIAL: NCT06029023
Title: Clinical And Radiographic Evaluation of Nano-Propolis, Nano-Curcumin and MTA as Direct Pulp Capping Agents in Young Permanant Teeth
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Collaborators: October 6 University (Other)
Responsible Party: Principal Investigator, Dalia Mohamed Elasser, Principal Investigator, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: october 6 university
Record Dates: First submitted 2023-07-22; First posted 2023-09-08 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Traumatic Pulp Exposure in Children
Keywords: MTA; PROPOLIS nano particles; nanocurcumin; dentin bridge; CBCT
MeSH Terms: interventions — mineral trioxide aggregate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- MTA (Active Comparator): Mineral trioxide aggregate MTA, The cement is made up of calcium, silicon and aluminium. The main constituent phases are tricalcium and dicalcium silicate and tricalcium aluminate.
  Interventions: Combination Product: MTA Cement, propolis nano particle, curcumin nanoparticles
- Nano propolis (Experimental): Propolis is a resinous substance that honey bees collect from different plant species. The most important pharmacologically active constituents in propolis are flavonoids, phenolics, and aromatics.
  Interventions: Combination Product: MTA Cement, propolis nano particle, curcumin nanoparticles
- Nano curcumin (Experimental): Curcumin (CUR), 7-bis (4-hydroxy-3-methoxyphenyl)-1,6- heptadien-3, 5-dione
  Interventions: Combination Product: MTA Cement, propolis nano particle, curcumin nanoparticles

INTERVENTIONS:
Combination Product: MTA Cement, propolis nano particle, curcumin nanoparticles — MTA or nano propolis or nano curcumin will then be placed over the remaining healthy pulp per the manufacturer's recommendation. The cavities will be lined with glass ionomer cement and a permanent composite restoration will be placed after 6 months. After treatment, a periapical radiograph and CBCT will be immediately taken with ultra-low dose The patients and their parents will be interviewed by telephone on day 1 and day 7 post-surgery about any pain or adverse reactions related to the treatment. Paracetamol will be prescribed if the patients had pain, however, no antibiotic will be used following the surgery. The patients will receive a 3-month follow-up clinical and periapical radiographic examination, together with 6 months clinical and CBCT examinations.

SUMMARY:
The aim of the study is to evaluate clinical and radiographic effect of nano propolis and nano curcumin as direct pulp capping agents in young permanent teeth.

.

DETAILED DESCRIPTION:
I. Materials:

1. Mineral trioxide aggregate (MTA)
2. Nano propolis
3. Nano curcumin
4. Glass ionomer

II. Methods:

Sample size calculation:

Sample size calculation was performed using G*Power version 3.1.9.7 based on the results of a previous study. The predicted sample size (n) was (54), i.e., 18 samples per group of the three groups, to detect results of dentin bridge thickness.

Sample preparation:

Patients will be recruited from the department of Pediatric Dentistry and Dental Public Heath, October 6 university. The study sample will be recruited among the children between 7 to 13 years old. The young permanent tooth eruption stage will be determined by the patient's age and radiographic evaluation before enrolling in the research study.

Before treatment, a periapical radiograph will be taken with ultra-low dose mode to assess the tooth radiographically for any sign of irreversible pulpitis.

Each tooth will be infiltrated with local anesthesia using 4% articaine with 1:100,000 epinephrine (Septanest, Septodont, France). The tooth will be isolated with a rubber dam and washed with 0.12% chlorhexidine. The cavity will be prepared, and the infected enamel and dentin will be removed with a round bur. The carious dentin close to the pulp will be removed using a spoon excavator. The pulp exposure position will be identified, and the inflamed pulp tissue (1.5-2 mm) will be gently removed using an abrasive diamond bur at high speed with copious sterilized normal saline. The remaining healthy pulp will be rinsed with 2.5% sodium hypochlorite, and moist, sterilized cotton pellets will be placed over the pulp stumps with light pressure for 2 min to achieve hemostasis. If the bleeding could not be controlled, the tooth will be excluded from this study. MTA or nano propolis or nano curcumin will then be placed over the remaining healthy pulp per the manufacturer's recommendation. To cover the exposure area, MTA and or nano propolis or nano curcumin will be placed using an amalgam carrier and non-toothed Adson forceps, respectively. The cavities will be lined with glass ionomer cement (Vitrebond, 3M ESPE, St. Paul, MN, USA), and a permanent composite restoration (Filtex Z350, 3M ESPE, Salt Lake City, UT, USA) will be placed after 6 months. After treatment, a periapical radiograph and CBCT (Planmeca. Romexis. Fenland) will be immediately taken with ultra-low dose mode (90 kVp, 5.6 mA, 4 × 5 cm FOV, and 0.2 vowel size) to serve as the baseline with a reduced dose, due to the need for future follow-ups.

The CBCT will be performed using an ultralow dose, small field of view, and appropriate radiation protection as described by the American Association of Endodontics (AAE) and the American Academy of Oral and Maxillofacial Radiology (AAOMR), and the European Society of Endodontology guidelines.

Shielding devices, a leaded thyroid collar, leaded glasses, and a leaded apron, will be used to protect the patient's thyroid gland, eye lens, body, respectively. The patients and their parents will be interviewed by telephone on day 1 and day 7 post-surgery about any pain or adverse reactions related to the treatment. Paracetamol will be prescribed if the patients had pain, however, no antibiotic will be used following the surgery. The patients will receive a 3-month follow-up clinical and periapical radiographic examination, together with 6 months clinical and CBCT examinations. The clinical and radiograph evaluations will be performed by blinded experienced endodontist and radiologist. The examiners will be trained in the evaluation criteria prior to the study. To determine the reliability of the evaluations, Kappa scores will be determined by the 2 examiners re-evaluating all cases 1 month after the initial evaluation performed. The intra- and inter-examiner Kappa scores of the clinical evaluation will be 1.0. For the radiographic evaluation, the intra-rater and inter-rater reliabilities will be 0.91 and 0.89, respectively. When there will be a disagreement, both examiners discussed the clinical and radiographic findings to achieve a consensus.

Variables:

Table 1: variables of the study:

Variables Referring to. Treatment agent MTA Nano propolis Nano curcumin

Time of assessment 6 months

Table 2: Interaction of variables of the study:

Variables Test MTA Nano propolis Nano curcumin Total Clinical examination 18 18 18 54 Dentin bridge formation. 18 18 18 54

Statistical Analysis:

All data will be collected, coded, tabulated and statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Young permanent teeth with deep carious lesions that led to a caries-exposed pulp after spoon excavation and a diagnosis of reversible pulpitis.
* The tooth has a pulp exposure caused by trauma that occurred within 48 h.

Exclusion Criteria:

* The patient has a history of systemic disease that interferes with pulp healing.
* The tooth has clinical signs and symptoms of irreversible pulpitis, e.g., spontaneous throbbing pain, tenderness to percussion, abnormal tooth mobility, swelling, or sinus tract.
* Radiographic evidence of internal or external resorption, inter-radicular bone loss, or periapical pathology.
* The tooth was non-restorable. During the study, if any symptoms of irreversible pulpitis, apical periodontitis, or infection occurred, the patients received the appropriate treatment following the institute protocol, including regenerative and root canal treatment.

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2022-12-20 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Incidence of pain or swelling | 1 week ,3 month , 6 month
  questionnaire applied for patient

SECONDARY OUTCOMES:
increase thickness of dentin bridge | baseline ,6 month
  digital cone beam radiograph

CONTACTS AND LOCATIONS:
Locations (1):
- Dalia Elasser, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No